CLINICAL TRIAL: NCT04010799
Title: A Phase Ib, Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Inhaled CHF 6333 After Single and Repeated Ascending Doses in Patients Affected by Cystic Fibrosis and Non Cystic Fibrosis Bronchiectasis
Brief Title: A Clinical Study to Investigate Safety, Tolerability and Distribution of CHF 6333 After One or After Repeated Inhalation in Patients With Cystic Fibrosis (CF) and in Patients With Non Cystic Fibrosis (NCFB) Bronchiectasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-06333AA1-16; 2018-002508-15 (EudraCT Number)
Record Dates: First submitted 2019-06-10; First posted 2019-07-08 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis; Non-Cystic Fibrosis Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Part I:
  Randomised, double-blind, placebo-controlled, single-dose escalation, cross-over design in one cohort of CF patients and in one cohort of NCFB patients.
  Part II:
  Randomised, double-blind, placebo-controlled, repeated-dose, parallel-group design in one cohort of CF patients and in one cohort of NCFB patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF6333 (Experimental): CHF6333 Active (part I - SAD). Once daily inhaled single dose of CHF6333 at each period (three dose level).
  CHF6333 Active (part II -MD). Once daily inhaled multiple dose of CHF6333 for 7 consecutive days.
  Interventions: Drug: CHF 6333
- CHF6333 Placebo (Placebo Comparator): Part I (SAD): Single dose of placebo matching CHF6333 at each period
  Part II (MD): Once daily multiple doses of placebo matching CHF6333 for 7 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF 6333 — CHF 6333 - Part I - SAD CHF 6333 - Part II - MD
  Arms: CHF6333
Drug: Placebo — Placebo - Part I - SAD Placebo Part II - MAD
  Arms: CHF6333 Placebo

SUMMARY:
CHF 6333 is a medicinal product on development for the treatment of cystic fibrosis and non-CF bronchiectasis and undergoing clinical testing. It has not yet been approved by the authorities for the treatment of these diseases.

CHF6333 is an inhaled anti-inflammatory which mechanism of action is based on the inhibition of Human Neutrofil Elastase.

The safety and tolerability of single and repeated ascending doses of inhaled CHF 6333 was previously investigated in healthy subjects: information was gathered on the uptake, distribution and excretion of the medicinal product being tested (pharmacokinetics). In this current clinical trial CHF 6333 will be tested in patients(CF and NCFB) for the first time.

Three dose level will be tested during the first part of the study, as single administration. One repeated dose will be administered in the second part of the study.

ELIGIBILITY:
INCLUSION CRITERIA:

CF patients:

* Patient's written informed consent obtained prior to any study-related procedure;
* Male or female patient ≥ 18 years old with a confirmed historical diagnosis of cystic fibrosis;
* Ability to provide a spontaneous sputum sample at screening;
* Non- or ex-smokers who smoked < 10 pack years and stopped smoking > 1 year before screening visit;
* Patient in stable clinical condition and free from exacerbation for at least 4 weeks prior to screening and/or prior to randomisation;
* Patient on stable concomitant treatment regimen within 4 weeks prior to screening and/or prior to randomisation;
* Patient with pre-bronchodilator FEV1 ≥ 50% of predicted normal at screening and/or prior to randomisation;
* Vital signs within normal limits at screening and prior to randomisation;

NCFB patients:

* Patient's written informed consent obtained prior to any study-related procedure;
* Male or female patient ≥ 18 years old with a diagnosis of Bronchiectasis confirmed by a historical Chest CT;
* Presence of clinically significant symptoms related to Bronchiectasis, such as daily cough that occurs over months or years, daily production of large amount of sputum, shortness of breath, wheezing chest pain;
* Ability to provide a spontaneous sputum sample at screening;
* Non- or ex-smokers who smoked < 10 pack years and stopped smoking > 1 year before screening visit;
* Patients in stable clinical condition and free from exacerbation since at least 4 weeks before screening and/or prior to randomisation;
* Patients on stable concomitant treatment regimen within 4 weeks prior to screening and/or prior to randomisation
* Patient with pre- bronchodilator FEV1 ≥ 50% of predicted normal at screening and/or prior randomization visit;
* Vital signs within normal limits at screening and prior to randomisation

EXCLUSION CRITERIA CF Patients

* Patient with BMI ≤ 17
* History of a clinically meaningful unstable or uncontrolled chronic comorbidity in the opinion of the Investigator;
* Unstable pulmonary status or symptomatic respiratory tract infection and related changes in therapy for pulmonary disease as per Investigator's judgment within 4 weeks before screening or prior to randomisation;
* Abnormal and clinically significant 12-lead ECG at screening or prior to randomisation;
* History of asthma based on objective evidence;
* History of malignancy, solid organ/haematological transplantation;
* Patient with evidence of active Nontuberculous Mycobacteria (NTM) and Tuberculous Mycobacteria (TM) infection or related bronchiectasis in the past 12 months;
* Patient with a positive test for active Allergic Bronchopulmonary Aspergillosis (ABPA) infection confirmed at screening or patient withABPA related bronchiectasis.
* Pregnant or lactating women.
* Patient on non-steroidal anti-inflammatory drugs (NSAIDs) within 4 weeks prior to screening or prior to randomization visit.
* Patient on cystic fibrosis transmembrane conductance regulator (CFTR) modulators and correctors if not on stable treatment regimen for at least 3 months prior to screening or prior to randomization.
* Positive HIV1 or HIV2 serology at screening; Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C at screening (i.e. positive HB surface antigen (HBsAg), HB core antibody (anti-HBc), HC antibody);

NCFB Patients

* Patient with BMI ≤ 17
* History of a clinically meaningful unstable or uncontrolled chronic comorbidity in the opinion of the Investigator;
* Unstable pulmonary status or symptomatic respiratory tract infection and related changes in therapy for pulmonary disease as per Investigator's judgment within 4 weeks before screening or prior to randomisation.
* Abnormal and clinically significant 12-lead ECG at screening or prior to randomisation that results in active medical problem which may impact the safety of the patients as per Investigator's judgment.
* History of malignancy, solid organ/haematological transplantation;
* Known diagnosis of cystic fibrosis. A negative sweat test is required at screening (sweat chloride should be < 40 mmol/L);
* History of asthma based on objective evidence of the condition;
* Patient with primary diagnosis of COPD in the opinion of theInvestigator;
* Patient with rheumatoid factor positivity;
* Patient with evidence of active Nontuberculous Mycobacteria (NTM) and Tuberculous Mycobacteria (TM) infection or related bronchiectasis in the past 12 months;
* Patient with a positive test for active Allergic Bronchopulmonary Aspergillosis (ABPA) infection confirmed at screening or patient with ABPA related bronchiectasis;
* Patient with Connective Tissue Disease (CTD) related bronchiectasis;
* Diagnosis of common variable immunodeficiency (CVID);
* Patient on any antibiotics (except for stable macrolides treatment),oral, inhaled and IV, within 4 weeks prior to screening or prior to randomisation;
* Patient on oral corticosteroids within 4 weeks prior to screening visit or prior to randomization.
* Patient on non-steroidal anti-inflammatory drugs (NSAIDs) within 4 weeks prior to screening or randomization visit.
* Patient on Carbocysteine and Mannitol treatment within 4 weeks before the screening or randomization visit.
* Patient with traction bronchiectasis;
* Patient with any condition that prevent them to use inhaledantibiotics (including patients who previously experienced adverse reaction to inhaled antibiotics;
* Patient treated with monoclonal antibodies (mAb);
* Pregnant or lactating women.
* Positive HIV1 or HIV2 serology at screening; Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C at screening (i.e. positive HB surface antigen (HBsAg), HBcore antibody (anti-HBc), HC antibody).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Adverse event | Part I: Baseline through end of treatment (up to a maximum of 30 days after last study drug intake) ; Part II Baseline through end of treatment (up to a maximum of 30 days after last study drug intake)
  Occurrence and severity of adverse events
Change in Vital signs | Part I: Day 1 pre-dose up to 6 hours post dose. Part II: Day 1 and Day 7 pre dose up to 6 hours post dose
  Change in Systolic and Diastolic blood pressure
Heart Rate | Part I: Day 1 pre dose up to 8 hours post dose. Part II: Day 1 and Day 7 pre dose up to 12 hours post dose
  Change in Heart Rate
PR interval | Part I: Day 1 pre dose up to 8 hours post dose. Part II: Day 1 and Day 7 pre dose up to 12 hours post dose
  Change in PR interval
QRS interval | Part I: Day 1 pre dose up to 8 hours post dose. Part II: Day 1 and Day 7 pre dose up to 12 hours post dose
  Change in QRS interval
QTCf interval | Part I: Day 1 pre dose up to 8 hours post dose. Part II: Day 1 and Day 7 pre dose up to 12 hours post dose
  Change in QTCf interval
FEV1 | Part I: Day 1 pre dose up to 6 hours post dose. Part II: Day 1 and Day 7 pre dose up to 6 hours post dose. Day 2 -6: pre dose up to 2 hours post dose
  Change in FEV1

SECONDARY OUTCOMES:
AUC | Part I: Day 1. Part II Day 1-7
  Area under the plasma concentration curve
Cmax | Part I: Day 1. Part II Day 1-7
  Peak plasma concentration
T max | Part I: Day 1. Part II Day 1-7
  Time to reach the maximum plasma concentration
C24h | Part II: Day 5 Day 6
  Trough drug concentration 24 h post dose
Rac | Part II: Day 7
  Accumulation ratio
NE activity | Part I: Day -1 Day 1. Part II: Day -1 - 7
  Change in neutrophil elastase activity in sputum

CONTACTS AND LOCATIONS:
Locations (1):
- IKF Institut für klinische Forschung Pneumologie, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No